CLINICAL TRIAL: NCT05438797
Title: Clinical Study on the Safety and Efficacy of Specific TIL-TCM Cells for Advanced Relapse-refractory or Metastatic Pancreatic Cancer
Brief Title: The Safety and Efficacy of Specific TIL-TCM Cells for Advanced Relapse-refractory or Metastatic Pancreatic Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sizhen Wang (Other)
Collaborators: Shanghai Biomed-union Biotechnology Co., Ltd. (Unknown)
Responsible Party: Sponsor-Investigator, Sizhen Wang, Clinical Study on the Safety and Efficacy of specific TIL-TCM cells for advanced relapse-refractory or metastatic pancreatic cancer, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022DZKY-039-02
Record Dates: First submitted 2022-06-26; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Advanced Pancreatic Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adoptive TIL-TCM transfer (Experimental): TIL-TCM cells are isolated from the patients' Tumor tissue (or ascites) and peripheral blood obtained before standard chemotherapy and then cultured ex-vivo. The first infusion will be conducted in 7-10 days after chemotherapy and is assessed by the investigators.TIL-TCM cells are transfused to patients in a dosage escalated manner.The total dose was 1× 109-1 ×1010 cells.After cell infusion, IL-2 was administered at 720000 IU/kg (based on whole body weight) by intravenous (I.V.),every 8 hours for up to 4 days.
  Interventions: Drug: Adoptive TIL-TCM transfer therapy

INTERVENTIONS:
Drug: Adoptive TIL-TCM transfer therapy — Abraxane:100-200 mg/m2，QD×1D;Cyclophosphamide:15-35 mg/kg/d，QD×2D. Biological: Adoptive TIL-TCM transfer therapy
  Other Names: TIL-TCM

SUMMARY:
Clinical Study on the Safety and Efficacy of specific TIL-TCM cells for advanced relapse-refractory or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
This is a single arm, open-label, single-center study.This study is indicated for advanced relapse-refractory or metastatic pancreatic cancer.The selections of dose levels and the number of subjects are based on clinical trials of similar foreign products. Primary objective is to explore the safety, main consideration is dose-related safety.

ELIGIBILITY:
Inclusion Criteria:

1. Aged≥18 years old and ≤70 years old when signing the informed consent; regardless of gender;Body weight>40kg.
2. Patients with advanced recurrent refractory or metastatic pancreatic cancer who have failed at least one standard treatment or who are unable to tolerate, unwilling or financially unable to receive standard treatment.
3. The subject will have at least one eligible tissue or sample available for cell preparation.
4. Patients with brain metastatic lesions who are asymptomatic , the diameter of a single lesion ≤1 cm, and the number of lesions ≤3 may be eligible.
5. Patients should have good clinical presentation status (ECOG 0 or 1).
6. HIV antibody and treponema pallidum antibody was negative.
7. Vital organ function test (do not accept any cytokines or blood transfusion within 14 days prior to test):

1)absolute neutrophil count (ANC) ≥1000/μL; 2)White blood cell count (WBC) 3000/μL; 3)Platelet count (PLT) 75,000 /μL; 4)Hemoglobin (Hb) > 8.0 g/dL; 5) Coagulation: activated partial thromboplastin time (APTT) ≤1.5×ULN, international normalized ratio (INR) or Prothrombin time (PT)≤1.5×ULN; 6) Liver functions: alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤5.0 ×ULN; 7) Liver functions:Total bilirubin (TBIL)<1.5×ULN (baseline value normal); <1.0 - 1.5×ULN( baseline value abnormal); If diagnosed as Gilbert syndrome, ≤3.0 mg/dL; The test results should prevail of the center laboratory ; 8)Renal function: eGFR>60 mL/min or 6-24 hours CrCl>60 mL/min; 9)Heart Doppler ultrasound:LVEF≥50%;

8.Non-surgically sterilized women of child-bearing age are required to consent to use at least one medically approved contraceptive method during the study and one year after completion.Women of child-bearing age must be negative for pregnancy test at 7 days before initiation of the treatment.Male subjects must agree to use medically approved contraception from the time they sign the informed consent form to the time they leave the study.

9.Expected survival no less than 3 months.

Exclusion Criteria:

1. Pregnancy or lactation;
2. Active infections requiring systemic anti-infective therapy ( topical antibiotics excepted);
3. Patients who are taking systemic steroids or immunosuppressive drugs;
4. Hepatitis B (hepatitis B surface antigen [HbsAg] and/or core antibody [HbcAb] positive, HBV-DNA<1000 copies /mL can be included);
5. Hepatitis C ( HCV antibody positive and HCV-RNA positive);
6. Serious autoimmune diseases or immunodeficiency disease, such as ulcerative colitis, Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus (SLE) and autoimmune vasculitis (eg., Wegener's granulomatosis);
7. Allergic:Severe allergies to the drugs used in the study; Contraindications for IL-2 used ;
8. Patients with other active malignancies within the past 5 years, but not those who were clinically cured within 5 years of diagnosis of cervical epithelial carcinoma, basal or squamous skin cancer, superficial bladder cancer, breast cancer in situ and did not require follow-up;
9. Any mental diseases, including dementia and changes in mental status that may influence the understanding about the informed consent and questionnaire;
10. Unstable disease of heart head blood-vessel, including but not limited to, the heart cerebrovascular accident or transient ischemic (within 6 months prior to screening) myocardial infarction (within 6 months prior to screening)/vein thrombosis (within 6 months prior to screening, require surgery to repair the aortic aneurysm or proximal artery thrombosis group shall not enter into) unstable angina New York Heart Association (NYHA) Classification≥ III congestive heart failure severe arrhythmias poorly controlled by medications and severe hypertension that cannot be controlled by treatment or is untreated (systolic pressure≥160 mmHg and/or diastolic pressure≥100 mmHg );
11. Patients with severe interstitial pneumonia other active pneumonia or bronchospasm and other respiratory diseases that seriously affect lung function;
12. Patients with active gastrointestinal bleeding;
13. Had major surgery within 1 month prior to screening or during the study ;
14. Enrolled in other clinical trials (including other adoptive cell immunotherapies) and used the investigational drug within 1 month prior to screening.
15. Have received live attenuated vaccine within 1 month prior to screening or are expected to receive live attenuated vaccine during the study ;
16. Received any systemic antitumor drug therapy (including chemotherapy, radiotherapy, molecular targeted therapy, immunotherapy or other biotherapy) within 4 weeks prior to pretreatment;
17. Have previously received allogeneic bone marrow transplantation or solid organ transplantation;
18. Alcohol, drug or substance abuse;
19. Judged as serious uncontrollable diseases by the researchers, or other conditions that may interfere with the treatment and therefore being ineligible.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2021-04-02 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days after TIL-TCM cells infusion
  To evaluate the Safety and Effectiveness of specific TIL-TCM cells in the Treatment of patients with advanced relapse-refractory or metastatic pancreatic cancer
Maximum Tolerated Dose（MTD） | Baseline up to 28 days after TIL-TCM cells infusion
  To evaluate the Safety and Effectiveness of specific TIL-TCM cells in the Treatment of patients with advanced relapse-refractory or metastatic pancreatic cancer
incidence of adverse events( AE )and Serious adverse events(SAE) | up to 72 weeks after TIL-TCM cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria.

SECONDARY OUTCOMES:
Overall response rate (ORR) | 18 months
  ORR is defined as the percentage of patients who have a clinical response (objective tumor regression).ORR is computed by: the sum of the number of patients with Complete Response (CR) and number of patients with Partial Response (PR) / total number of patients. The total number of patients is the sum of the number of patients with CR, PR, stable disease (SD) or progressive disease (PD). The Response Evaluation Criteria in Solid Tumors (RECIST v1.1) is used as the criteria to determine whether a tumor disappears (CR), shrinks (PR), stays the same (SD) or gets bigger (PD).
Duration of response (DOR) | 18 months
  DOR is the time between the initial response to treatment per RECIST v1.1 and subsequent disease progression among patients achieving Complete Response (CR) or Partial Response (PR). RECIST v1.1 is used as the criteria to determine whether a tumor disappears (CR) or shrinks (PR).
Progression-free survival (PFS) | 18 months
  PFS is the length of time from the date patient enrolled in to the date on which tumor progresses or the patient dies for any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Xinbo Wang, MD, Study Director — Jinling Hospital,Nanjing University
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China